CLINICAL TRIAL: NCT03311230
Title: Social Incentives To Encourage Physical Activity and Understand Predictors
Acronym: STEPUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Deloitte (Industry)
Responsible Party: Principal Investigator, Mitesh Patel, Mitesh S. Patel, Director, Penn Medicine Nudge Unit, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 827508
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants in this arm will receive no other interventions during the 9 month study period
- Supportive social incentive (Experimental): Participants will identify a family member or friend to support them during a gamification intervention.
  Interventions: Behavioral: Supportive social incentive
- Competitive social incentive (Experimental): Participants will compete in a gamification intervention in groups of three.
  Interventions: Behavioral: Competitive social incentive
- Collaborative social incentive (Experimental): Participants will collaborate in groups of three in a gamification intervention
  Interventions: Behavioral: Collaborative social incentive

INTERVENTIONS:
Behavioral: Supportive social incentive — A family member or friend will be used as a support person in this study, to receive updates and support the participant in their progress.
  Arms: Supportive social incentive
Behavioral: Competitive social incentive — Participants in this intervention will be competing against each other in the game.
  Arms: Competitive social incentive
Behavioral: Collaborative social incentive — Participants in this intervention will be working with each other in the game.
  Arms: Collaborative social incentive

SUMMARY:
This study tests the effectiveness of three social incentive-based gamification interventions to increase physical activity using a 24-week intervention period with a 12-week follow-up.

DETAILED DESCRIPTION:
This is a four-arm randomized, controlled trial with a 24-week intervention period and 12-week follow-up period. Participants are considered ready to be randomized once they have completed all surveys, established a baseline step count, and selected a step goal increase.Participants in the control arm will receive no other interventions during the 24-week intervention period or the 12-week follow-up period. Participants randomized to the one of the three intervention arms will have a 4-week ramp up towards their step goal. The participant will then be asked to maintain their goal during the 20-week "maintenance period" and the 12-week "follow-up period." Participants in arms 2-4 will be entered into an intervention approach that has points and levels designed to incorporate insights from behavioral economics. Participants in the supportive social incentive arm will be asked to identify a family member or friend to be their support sponsor. This sponsor will be encouraged to support the participant in their progress during the study. Participants in the competitive social incentive arm will be in a group of three total participants.At the end of each week the participants will receive notification that ranks them on their cumulative points in the study thus far and also displays their level.This feedback may help to induce participants to compete for the top spot among the group. Participants in the collaborative social incentive arm will be in a group of three total participants as a team. Each day one of the members of the group will be randomly selected to represent their team for that day. In this design, each person is accountable to the others on the team and this may induce a collaborative effort to meet their daily goals.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. ability to read and provide informed consent to participate in the study;
3. Self-reported body mass index (BMI) of 25 or greater.
4. Smartphone or tablet compatible with application for the wearable activity tracking device.

Exclusion Criteria:

1. Conditions that would make participation infeasible such as inability to provide informed consent, illiteracy or inability to speak, read, and write English;
2. conditions that would make participation unsafe such as pregnancy or being told by a physician not to exercise;
3. already enrolled in another study targeting physical activity;
4. any other medical conditions or reasons he or she is unable to participate in a physical activity study for 36 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewey J, Murphy S, Zhang D, Putt ME, Elovitz MA, Riis V, Patel MS, Levine LD. Effectiveness of a Text-Based Gamification Intervention to Improve Physical Activity Among Postpartum Individuals With Hypertensive Disorders of Pregnancy: A Randomized Clinical Trial. JAMA Cardiol. 2022 Jun 1;7(6):591-599. doi: 10.1001/jamacardio.2022.0553. PMID 35442393
- [Derived] Rewley J, Guszcza J, Dierst-Davies R, Steier D, Szwartz G, Patel M. Loss Aversion Explains Physical Activity Changes in a Behavioral Gamification Trial. Games Health J. 2021 Dec;10(6):430-436. doi: 10.1089/g4h.2021.0130. PMID 34860130
- [Derived] Patel MS, Small DS, Harrison JD, Fortunato MP, Oon AL, Rareshide CAL, Reh G, Szwartz G, Guszcza J, Steier D, Kalra P, Hilbert V. Effectiveness of Behaviorally Designed Gamification Interventions With Social Incentives for Increasing Physical Activity Among Overweight and Obese Adults Across the United States: The STEP UP Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1624-1632. doi: 10.1001/jamainternmed.2019.3505. PMID 31498375
- [Derived] Harrison JD, Jones JM, Small DS, Rareshide CAL, Szwartz G, Steier D, Guszcza J, Kalra P, Torio B, Reh G, Hilbert V, Patel MS. Social incentives to encourage physical activity and understand predictors (STEP UP): Design and rationale of a randomized trial among overweight and obese adults across the United States. Contemp Clin Trials. 2019 May;80:55-60. doi: 10.1016/j.cct.2019.04.001. Epub 2019 Apr 4. PMID 30954675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
Started | 151 | 151 | 150 | 150
Completed | 150 | 146 | 148 | 143
Not Completed | 1 | 5 | 2 | 7
Not completed — Withdrawal by Subject | 1 | 4 | 2 | 7
Not completed — Unrelated injury | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive | Total
Number analyzed (Participants) | 151 | 151 | 150 | 150 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.9) | 39.4 (10.1) | 38.7 (10) | 38.3 (10) | 38.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 41 | 37 | 43 | 175
  Male | 97 | 110 | 113 | 107 | 427
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White non-Hispanic | 72 | 72 | 80 | 81 | 305
  Black non-Hispanic | 10 | 9 | 8 | 5 | 32
  Asian non-Hispanic | 49 | 57 | 52 | 48 | 206
  Hispanic | 10 | 7 | 3 | 7 | 27
  Other | 10 | 6 | 7 | 9 | 32
Education level [Count of Participants; unit: Participants]
  High school graduate | 1 | 0 | 1 | 1 | 3
  Some college or specialized training | 8 | 5 | 6 | 4 | 23
  College graduate | 142 | 146 | 143 | 145 | 576
Marital status [Count of Participants; unit: Participants]
  Single | 43 | 31 | 38 | 39 | 151
  Married | 102 | 113 | 101 | 102 | 418
  Other | 6 | 7 | 11 | 9 | 33
Annual household income [Count of Participants; unit: Participants]
  < 50,000 | 1 | 1 | 1 | 2 | 5
  50,000 - 100,000 | 33 | 29 | 36 | 26 | 124
  > 100,000 | 117 | 121 | 113 | 122 | 473
Self-reported measures, health status [Count of Participants; unit: Participants]
  Excellent | 6 | 8 | 11 | 5 | 30
  Very good | 43 | 54 | 55 | 46 | 198
  Good | 84 | 63 | 66 | 69 | 282
  Fair | 16 | 22 | 18 | 28 | 84
  Poor | 2 | 4 | 0 | 2 | 8
Prior wearable device use [Count of Participants; unit: Participants] | 89 | 100 | 101 | 94 | 384
BMI, Mean (SD) [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (4.1) | 29.2 (4.8) | 29.7 (4.9) | 30.1 (5.7) | 29.7 (4.9)
Diabetes [Count of Participants; unit: Participants] | 10 | 4 | 5 | 11 | 30
Hyperlipidemia [Count of Participants; unit: Participants] | 27 | 22 | 27 | 29 | 105
Hypertension [Count of Participants; unit: Participants] | 23 | 16 | 17 | 20 | 76
Smoking actively [Count of Participants; unit: Participants] | 5 | 5 | 5 | 7 | 22
Baseline step count, Mean (SD) [Mean (Standard Deviation); unit: steps/day] | 6086 (2631) | 6297 (2571) | 6313 (2812) | 6120 (2583) | 6204 (2646)
Step goal selection, No. (%) [Count of Participants; unit: Participants]
  33% Increase from baseline | 64 | 56 | 60 | 56 | 236
  40% Increase from baseline | 19 | 14 | 20 | 24 | 77
  50% Increase from baseline | 19 | 31 | 22 | 32 | 104
  Custom goal at least 1500 steps > than baseline | 49 | 50 | 48 | 38 | 185
Step goal increase from baseline, mean (SD) [Mean (Standard Deviation); unit: steps/day] | 2144 (1160) | 2243 (923) | 2210 (1529) | 2200 (980) | 2199 (1169)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Steps
Description: Change in mean daily steps from baseline to main intervention period
Time Frame: weeks 5 to 24 of the intervention
Measure: Mean (Standard Deviation); unit: Steps/Day
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
Number analyzed (Participants) | 151 | 151 | 150 | 150
Steps/Day | 6162 (2142) | 6975 (2403) | 7237 (2934) | 6814 (2197)

2. Secondary Outcome: Change in Mean Daily Steps
Description: Change in mean daily steps from baseline through the follow-up period
Time Frame: Weeks 25 to 36 of the follow-up period
Measure: Mean (Standard Deviation); unit: Steps/Day
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
Number analyzed (Participants) | 151 | 151 | 150 | 150
Steps/Day | 5899 (2128) | 6432 (2320) | 6592 (2685) | 6038 (1640)

3. Secondary Outcome: Proportion of Participant-days That Step Goals Are Achieved
Description: proportion of days participants meet their step goal
Time Frame: Weeks 5 to 24 of the main intervention period.
Measure: Number; unit: Proportion of participant-days
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
Number analyzed (Participants) | 151 | 151 | 150 | 150
Proportion of participant-days | 0.25 | 0.36 | 0.41 | 0.36

4. Secondary Outcome: Proportion of Participant-days That Step Goals Are Achieved
Description: proportion of days participants meet their step goal
Time Frame: Weeks 25 to 36 of the follow-up period.
Measure: Number; unit: Proportion of participant-days
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
Number analyzed (Participants) | 151 | 151 | 150 | 150
Proportion of participant-days | 0.23 | 0.28 | 0.30 | 0.26

ADVERSE EVENTS:
Time Frame: Adverse event data was collected when participants were started in the study through the maintenance and follow-up periods (9 months, or 252 days).
Description: Mortality was not a risk associated with participation in our study.
Arm/Group | Control | Supportive Social Incentive | Competitive Social Incentive | Collaborative Social Incentive
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/151 | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/151 | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/151 | 1/151 | 0/150 | 0/150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=151) | Supportive Social Incentive (N=151) | Competitive Social Incentive (N=150) | Collaborative Social Incentive (N=150)
Broken foot (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — The participant suffered a broken foot and required surgery to repair.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT03311230/Prot_SAP_000.pdf